CLINICAL TRIAL: NCT05628090
Title: A retrosPective Descriptive Analysis Assessing the trEatment peRsistence to baSal InSulin in Type 2 diabEtes patieNTs in a Structured Patient Education Program in India
Brief Title: A Study of an Existing Database to Assess the Treatment Persistence to Basal Insulin in Type 2 Diabetes Mellitus Patients in a Structured Patient Education Program in India
Acronym: PERSISTENT
Status: Completed | Type: Observational
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Other Study IDs: LANTUL09644; U1111-1280-5131 (Registry Identifier: ICTRP); PDE0043 (Other: Sanofi Identifier)
Record Dates: First submitted 2022-11-16; First posted 2022-11-28 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2024-03

CONDITIONS: Type 2 Diabetes Mellitus (T2DM)
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study is to analyze data from an existing database named SAATH-7 Star, in order to assess the treatment persistence to basal insulin in Type 2 diabetes patients who had been enrolled in the SAATH-7 Star structured patient education program in India.

DETAILED DESCRIPTION:
This retrospective study will involve secondary analysis of already existing data of Indian T2DM patients who were administered subcutaneous injectable solutions of insulin glargine (Lantus® or Toujeo®), as per routine clinical practice and who were enrolled in a structured educational program named SAATH-7 Star. Six-months data for eligible patients, who were enrolled in the SAATH-7 Star Program during the index period of March 2019-August 2019, collected from the SAATH-7 Star database will be analyzed for the defined objectives. The index date is defined as the date of enrollment in SAATH-7 Star program i.e. 1st month, which will also be considered as the 'Baseline'

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged ≥ 18 years
* T2DM patients enrolled in SAATH-7 Star program during the index period from March 2019 to August 2019

Exclusion Criteria:

* Type 1 diabetes patients
* Patients with gestational diabetes

The above information is not intended to contain all considerations relevant to a potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Data will be analyzed for all T2DM patients ≥ 18 years of age, enrolled in the SAATH-7 Star program from March 2019 to August 2019, with a treatment length of 6 months.
Sampling Method: Non-Probability Sample
Enrollment: 47885 (Actual)
Dates: Start 2022-11-30 (Actual); Primary Completion 2023-12-29 (Actual); Study Completion 2023-12-29 (Actual)

PRIMARY OUTCOMES:
Proportion of patients persisting on insulin glargine (Lantus® or Toujeo®) at the end of 6th month | Month 6

SECONDARY OUTCOMES:
Proportion of patients persisting on insulin glargine (Lantus® or Toujeo®) at the end of 3rd month | Month 3
Proportion of patients persisting on Lantus® at the end of 3rd and 6th months | Month 3 and 6
Proportion of patients persisting on Toujeo® at the end of 3rd and 6th months | Month 3 and 6
Change in Lantus® dose at the end of 3rd and 6th months | Month 3 and 6
Change in Toujeo® dose at the end of 3rd and 6th months | Month 3 and 6
Proportion of patients on Lantus® who switched to other therapy at the end of 6th month | Month 6
Proportion of patients on Toujeo® who switched to other therapy at the end of 6th month | Month 6

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (1):
- Investigational Site Number :, Chilly-Mazarin, France

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org